CLINICAL TRIAL: NCT05258461
Title: An Innovative Smartphone Application for Adverse Event Management During Breast Cancer Adjuvant Chemotherapy: a Randomized Controlled Trial
Brief Title: An Innovative Smartphone Application for Adverse Event Management During Breast Cancer Adjuvant Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Smart
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: Application; Adverse Event; Quality of Life; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group will receive conventional adverse event management and have access to the smartphone app during chemotherapy.
  Interventions: Other: use of a smartphone app for adverse event management; Other: conventional adverse event management
- The control group (Active Comparator): The control group will receive conventional adverse event management during chemotherapy. Chemotherapy-related adverse events in the control group will be managed with symptomatic treatment, dietary and lifestyle prescription according to the doctors' clinical experience.
  Interventions: Other: conventional adverse event management

INTERVENTIONS:
Other: use of a smartphone app for adverse event management — At their enrollment, patients will receive detailed introduction and adequate assistance on the use of the smartphone app. The smartphone app will offer proper advice for adverse event management based on calculated results by artificial intelligence on the innovative app, which was developed by YL et al. It was specifically intended for risk prediction, early prevention, as well as management of symptoms and concerns during adjuvant chemotherapy in the treatment of breast cancer. The app consisted of 4 modules: (1) Module 1: clinical data collection. (2) Module 2: risk evaluation for 12 common adverse events during breast cancer chemotherapy. (3) Module 3: personalized prophylaxis based on predicted risks of adverse events. (4) Module 4: Q&A platform.
  Arms: The intervention group
Other: conventional adverse event management — Chemotherapy-related adverse events in the control group will be managed with symptomatic treatment, dietary and lifestyle prescription according to the doctors' clinical experience. For example, colony-stimulating factors and antibiotics may be used for febrile neutropenia, loperamide (or diphenoxylate plus atropine) as prophylaxis for diarrhea, together with eating low-lactose and low-fat frequent small meals. 5-hydroxytryptamine 3 receptor antagonist, neurokinin 1 receptor antagonist, and/or dexamethasone would be prescribed for patients at high risks of vomiting.

SUMMARY:
The aim of this study is to evaluate benefits of the app in breast cancer patients receiving the docetaxel, doxorubicin, and cyclophosphamide (TAC) chemotherapy. The investigators hypothesized that the addition of the app to conventional adverse event management would increase quality of life (QoL) scores and reduce adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. pathological diagnosis of invasive breast cancer
2. breast surgery within the past 2-8 weeks
3. adult female
4. must be able to use mobile phones
5. speak and write Chinese fluently to sign the informed consent

Exclusion Criteria:

1. severe comorbidity that interferes with outcome evaluation
2. insufficient Chinese language skills
3. inability to use mobile phones
4. cognitive disability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-10-07 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline quality of life scores at 4 months | 1 day before the first cycle, and 4 months after the first cycle (each cycle is 21 days)
  Quality of life scores will be assessed using the simplified Chinese version of the Organization for Research and Treatment of Cancer (EORTC QLQ-C30, version 3).

SECONDARY OUTCOMES:
Incidence and severity of 12 common adverse events | 4 months after the first cycle (each cycle is 21 days)
  The incidence and severity of 12 common adverse events will be measured with the WHO-toxicity scale.

OTHER OUTCOMES:
Login times | Documented automatically by the application every two weeks
  Login times to the application during chemotherapy
Average time spent on the application | Documented automatically by the application every two weeks
  Average time spent on the application each time
Questions addressed on the Q&A platform | Documented automatically by the application every two weeks
  Questions addressed on the Q&A platform

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Doctor, Study Director — Department of Breast Surgery, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No
The data will not become available to public.

REFERENCES:
- [Background] Cheng JX, Liu BL, Zhang X, Zhang YQ, Lin W, Wang R, Zhang YQ, Zhang HY, Xie L, Huo JL. The validation of the standard Chinese version of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) in pre-operative patients with brain tumor in China. BMC Med Res Methodol. 2011 Apr 22;11:56. doi: 10.1186/1471-2288-11-56. PMID 21513533
- [Background] Wan C, Meng Q, Yang Z, Tu X, Feng C, Tang X, Zhang C. Validation of the simplified Chinese version of EORTC QLQ-C30 from the measurements of five types of inpatients with cancer. Ann Oncol. 2008 Dec;19(12):2053-60. doi: 10.1093/annonc/mdn417. Epub 2008 Jul 24. PMID 18653703
- See also: WHO-toxicity scale — https://doi.org/10.1007/978-3-211-89836-9_1474
- See also: Guidelines of Chinese Society of Clinical Oncology (CSCO) on Diagnosis and Treatment of Breast Cancer (2020 version) — https://tbcr.amegroups.com/article/view/45555
- See also: (NCCN) Clinical Practice Guidelines in Oncology. Breast Cancer, Version 1.2022 — https://www.nccn.org/